CLINICAL TRIAL: NCT02184299
Title: A Multicenter, Randomized, Open-label, Controlled Study of Nevirapine (VIRAMUNE®) and a Short Course of Prednisone to Determine the Safety and Effectiveness of This Strategy in Preventing Nevirapine (VIRAMUNE®) Associated Rash.
Brief Title: Study of Nevirapine and Prednisone to Determine the Safety and Effectiveness in Preventing Nevirapine Associated Rash in Human Immunodeficiency Virus (HIV) Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1286
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Prednisone

ARMS (2):
- Nevirapine + Prednisone (Experimental): week 1-2: Nevirapine + Prednisone
  week 3-24: Nevirapine alone
  Interventions: Drug: Nevirapine; Drug: Prednisone
- Nevirapine (Active Comparator): week 1-24: Nevirapine
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: Nevirapine
Drug: Prednisone
  Arms: Nevirapine + Prednisone

SUMMARY:
Study to determine the incidence of rash between the group receiving nevirapine without prednisone and the group receiving nevirapine with prednisone

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of any ethnic group between the ages of 18 and 65 years of age

  * Women of childbearing potential had to utilize adequate birth control to prevent pregnancy for study duration. Due to possibility that study drugs could alter the effectiveness of oral contraceptives or depo-progesterone, oral contraceptives or depo-progesterone were not to be used as the sole form of birth control for the duration of this study
  * Women of childbearing potential had to have a negative serum human chorionic gonadotropin (b-hCG) within 14 days prior to initiation of study therapy
* Presence of HIV-1 infection as documented by any licensed Enzyme-Linked Immunosorbent Assay (ELISA) test kit and confirmed by either Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA at any time prior to study entry
* A CD4+ cell count of 100 cells/mm³ documented within 30 days of baseline visit. If a patient had a history of a clinical AIDS defining event, i.e. Pneumocystis carinii pneumonia (PCP), Kaposi sarcoma, etc, his/her CD4+ cell count had to be >= 200 cells/mm³
* Patients could have either a) no prior antiretroviral therapy or b) prior antiretroviral therapy but no Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTI) therapy. Antiretroviral experienced patients eligible to enroll in this study were patients who had any of the following characteristics

  * Switching Patients: Patients with two consecutive ultra-sensitive HIV-RNA assay results below the limit of quantification (BLQ) at least one week apart
  * Patients Optimizing Therapy: Patients who had responded with substantial drops in HIV-RNA counts without reaching BLQ or patients who had failed their current regimen and needed to change to a new drug regimen
  * Patients Re-starting Therapy: Patients who were antiretroviral experienced but had not received antiretroviral therapy in the previous three months before enrolling in this study All antiretroviral experienced patients had to have been on a stable regimen or for at least three months immediately prior to their enrollment or they had to have been on no antiretroviral therapy for at least three months immediately prior to their enrollment
* Ability and willingness to give written informed consent and comply with study requirements
* Patients must have had an ambulatory performance score of >= 80 on the Karnofsky scale

Exclusion Criteria:

* Female patients who were pregnant or breast-feeding
* Patients with an acute and/or active AIDS defining illness
* History of any illness or drug allergy that in the opinion of the Investigator could confound the results of the study or pose additional risk in administering nevirapine to the patient
* Patients with active invasive infections including pneumonia, septicemia, meningitis and encephalitis; not including upper respiratory infections, dermatologic infection, oral infection and urinary tract infection
* Patients who where currently taking any prescription or non-prescription drug that in the opinion of the investigator in consultation with Boehringer Ingelheim Pharmaceuticals Incorporated (BIPI) medical monitor could interfere with either the absorption, distribution or metabolism of nevirapine or prednisone
* The following laboratory parameters documented within 30 days prior to baseline visit:

  * Hemoglobin < 9.1 g/dL for men; < 8.9 g/dL for women
  * Absolute neutrophil counts < 750 cells/mm³
  * Platelet counts < 50000 platelets/mm³
  * AST (SGOT)/ALT (SGPT) > five times upper limit of normal range (ULN)
  * Creatinine > two times ULN
* Documented or suspected acute hepatitis within 30 days prior to baseline visit irrespective of Aspartate Aminotransferase (AST) Serum Glutamic-Oxaloacetic Transaminase (SGOT) and Alanine Aminotransferase (ALT) Serum Glutamic-Pyruvic Transaminase (SGPT) values that were five times ULN
* Unexplained temperature > 38.5 °C for any seven days or chronic diarrhea defined as more than three stools per day that persisted for 15 days within 30 days prior to baseline visit
* History of illnesses that contraindicated the use of prednisone such as hypertension, diabetes and diseases of the adreno-pituitary axis. Any chronic gastrointestinal conditions that could interfere with study drug absorption
* Receipt of the following

  * Any NNRTI therapy at anytime prior to baseline visit
  * Interferons, interleukins or any vaccine including HIV vaccine within 30 days prior to baseline visit
  * Any investigational agents that needed to be continued during the study
  * Abacavir
  * Patients who would be taking known inhibitors or inducers of P450 metabolic enzymes including ketoconazole, itraconazole, rifampin and phenytoin were not enrolled. In addition the following drugs were not allowed during the study: cytochrome P450 3A4 substrates such a terfenadine, astemizole, cisapride, triazolam and midazolam. Non-nucleoside reverse transcriptase inhibitors other than study-provided nevirapine were not allowed
* The presence of skin rash or mucosal lesions that in the opinion of the Investigator could compromise the wellbeing of the patient or confound that assessment of a nevirapine-associated rash. Localized skin rashes (e.g. facial folliculitis or contact dermatitis) were not to be the only basis for exclusion from this trial
* Presence of occult (microscopic) or frank (macroscopic) blood in the stools
* Any medical condition which in the opinion of the Investigators would interfere with the patient's ability to participate in or adhere to the requirements of this protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 1999-04; Primary Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
Incidence of rash | up to 42 days after initiation of nevirapine

SECONDARY OUTCOMES:
Severity of rash | up to 42 days after initiation of nevirapine
Change in Human Immunodeficiency Virus -1 Ribonucleic Acid (HIV-1 RNA) count | up to 24 weeks
Number of patients with adverse events | up to 198 days
Change in Lymphocytes expressing CD4+ Surface Marker (CD4+) count | up to 24 weeks